CLINICAL TRIAL: NCT02487667
Title: Effects of a Therapeutic Exercise Program by a Feedback a Motor Control System in the Elderly
Brief Title: Therapeutic Exercise Training in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Alazne Ruiz de Escudero Zapico, Physical Therapist, Universidad de Zaragoza
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A14/001
Record Dates: First submitted 2015-06-22; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Functional Insufficiency; Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Active Comparator): Therapeutic exercise
  Interventions: Device: Therapeutic exercise by fitness machines
- Control Group (No Intervention): No treatment

INTERVENTIONS:
Device: Therapeutic exercise by fitness machines — Therapeutic exercise program by using 8 exercise machine circuit
  Arms: Intervention Group

SUMMARY:
In adulthood, limited mobility and pain are very common and often the first clear sign of functional decline. The loss of independent mobility is related to higher rates of functional disability and mortality; however, it is also susceptible to interventions through exercises. With aging, changes in peripheral and central nervous system also occur, which lead to degradation of the sensory receptors as well as a loss of muscle mass and coordination. However, both, structural and functional dysfunctions of the nervous system, can be mitigated by increasing physical activity.

The aim of this study is therefore, to study the effects on pain and functional capacity of a therapeutic exercise training program in an adult people sample. The therapeutic exercise machines proposed in this trial have not been previously analyzed and provide insight into this field due to their design. The design of this new machines allows the adaptation to each concrete clinical situation by the adjustment of different parameters such as feedback, range of movement, time of repetition, intensity, speed and rhythm, which facilitate motor control training.

ELIGIBILITY:
Inclusion Criteria:

* Ability to complete self-reported questionnaires
* Autonomous ambulation that allows the realization of functional test
* Accept and consent to voluntarily participate in the study
* Preclinical mobility restriction and/or pain in absence of important pathologies.

Exclusion Criteria:

* Present contraindications for physical exercise
* Receiving physiotherapy treatment during the time of the trial.
* Modification of physical habits
* Change the pattern or usual pharmacotherapy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain intensity | 8 weeks
  Measured by Visual Analogue Scale
Change from baseline in range of movement | 8 weeks
  Measured by a motion capture system

SECONDARY OUTCOMES:
Body composition | 8 weeks
  weight, BMI
Functional capacity | 8 weeks
  spirometry and functional tests of the extremities
Quality of life | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alazne Ruiz de Escudero Zapico, Principal Investigator — Unidad de Investigacion en Fisioterapia. Universida de Zaragoza
Locations (1):
- Alazne Ruiz de Escudero Zapico, Zaragoza, Zaragoza, Spain